CLINICAL TRIAL: NCT01308619
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Evaluation of Rosacea-related Inflammatory Biochemical Markers in the Skin of Adults With Papulopustular Rosacea Treated With Daily Doxycycline 40 mg (30 mg Immediate Release / 10 mg Delayed Release Beads) Capsules
Brief Title: Evaluation of Rosacea-related Inflammatory Biochemical Markers in Adult Skin When Treated With Oracea® vs Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: US10150
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2014-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oracea® (Active Comparator): Doxycycline 40 mg (30 mg immediate release / 10 mg delayed release beads) Capsules
  Interventions: Drug: Doxycycline
- placebo (Active Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Doxycycline — doxycycline 40 mg (30 mg immediate release / 10 mg delayed release beads) Capsules, oral, one capsule daily in the morning
  Other Names: Oracea®
  Arms: Oracea®
Other: Placebo — Placebo, oral, one capsule daily in the morning
  Arms: placebo

SUMMARY:
The objective of this study is to determine the clinical effects of doxycycline 40 mg (30 mg immediate release and 10 mg delayed release beads) capsules (Oracea®) as compared to placebo in the skin of adults with papulopustular rosacea and to identify a correlation, if any, with rosacea-related inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female aged 18 to 70 years inclusive
* Subject with papulopustular rosacea (5 to 40 papules or pustules)

Exclusion Criteria:

* Subject has any other active dermatological condition on face that may interfere with the conduct of the study
* Subject uses proton pump inhibitors for treatment of gastroesophageal reflux within 30 days prior to baseline visit or during the study
* Subject uses spironolactone within 30 days prior to baseline visit or during the study
* Subject requires chronic treatment (>14 days) with sulfa drugs, erythromycin, cephalosporins and quinolones within 30 days prior to baseline visit or during the study
* Subject has used tetracycline antibiotics within 30 days prior to baseline visit or during the study
* Subject has used penicillin antibiotics within 30 days prior to baseline visit or during the study
* Subject uses topical or oral dapsone
* Subject has had a change in hormonal therapy within 3 months of initiation of therapy or during the study
* Subject has used systemic immunosuppressants (e.g. corticosteroids, cyclosporine, imuran, biologics, mycophenolate mofetil) within 30 days prior to baseline visit. For subjects who have received treatment with biologics, treatment must have been discontinued within 90 days prior to baseline
* Subject has used any systemic therapy directed at improving rosacea, including antibiotics, within 30 days prior to baseline visit
* Subject has used systemic retinoids within 6 months of the baseline visit
* Subject takes niacin at a dosage of 500 mg or more per day
* Subject has used any topical rosacea therapy including topical antibiotics, topical retinoids, topical sodium sulfacetamide preparations, topical benzoyl peroxides, topical vasoconstricting agents (e.g., oxymetazoline) topical calcineurin inhibitors (e.g. tacrolimus, pimecrolimus) within 30 days prior to baseline visit
* Subject has been treated with another investigational drug or device within 30 days of baseline visit. For subjects who received experimental biologic treatment, treatment must have been discontinued within five half lives of the baseline visit.
* Subject has a known allergy to any of the components of the study products, and/or a known hypersensitivity to tetracyclines
* Subject is using a clinically significant concomitant drug (e.g., use of long term non-steroidal anti-inflammatory agents unless used only on a PRN basis less than 7 days per month)
* Subject has used vasodilators or an adrenergic blocking agent within 6 weeks of baseline visit (except subjects on stable dose for greater than 3 months)
* Subject has had laser or light therapy on the face within 3 months of the baseline visit
* Subject with active ocular rosacea and/or blepharitis/meibomianitis requiring systemic treatment by an ophthalmologist
* Subject with rhinophymatous rosacea
* Subject with a history of noncompliance with a treatment regimen
* Subject is at risk in terms of precautions, warnings, and contraindications (see package insert)
* Subject has previously failed to have improvement of rosacea with appropriate use of systemic tetracycline family of antibiotics
* Subjects with a recent history of alcohol and/or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (10):
- United States (10):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Therapeutics Clinical Research, San Diego, California
  - Hudson Dermatology, Evansville, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Michigan Center for Research Corp, Clinton Township, Michigan
  - Skin Search of Rochester, Inc, Rochester, New York
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Derm Research, Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 9 May 2011, last subject last visit 2 July 2012
Groups:
- Oracea®: Doxycycline 40 mg (30 mg immediate release / 10 mg delayed release beads) Capsules for 12 weeks
- Placebo Capsules: Placebo capsules for 12 weeks
Period: Overall Study
Arm/Group | Oracea® | Placebo Capsules
Started | 84 | 86
Completed | 77 | 83
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oracea® | Placebo | Total
Number analyzed (Participants) | 84 | 86 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (11.4) | 48.7 (10.8) | 49.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 60 | 121
  Male | 23 | 26 | 49
Region of Enrollment [Number; unit: participants]
  United States | 84 | 86 | 170

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Inflammatory Lesion Counts
Description: Mean change in inflammatory lesion counts from baseline to week 12
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: inflammatory lesions
Arm/Group | Oracea® | Placebo
Number analyzed (Participants) | 84 | 86
inflammatory lesions | -4.3 (7.9) | -3.2 (8.6)

2. Secondary Outcome: Change From Baseline in Biochemical Markers of Rosacea From Tape Stripping and/or Skin Biopsy From Baseline to Week 12
Description: Mean change from baseline to week 12 in biochemical markers of rosacea and expression in skin samples. A biological marker is a substance used as an indicator of a biological state such as rosacea. Biochemical markers are serine protease activity and expression, metalloprotease activity and expression, and production of leucine leucine-37 [LL-37] peptide.
Time Frame: baseline to week 12
Population: Treatment success was defined as all subjects from either treatment group with a score of clear or near clear on the Investigator's Global Assessment (IGA) scale. Treatment failure was defined as all subjects from either treatment group with a score of mild, moderate, or severe on the IGA scale.
Measure: Mean (Standard Deviation); unit: micr grams protein
Arm/Group | Treatment Success | Treatment Failure
Number analyzed (Participants) | 49 | 111
micr grams protein
  Cathelicidin | -0.0931 (0.5491) | -0.0379 (0.1545)
  KLK5 | -0.0034 (0.0110) | -0.0049 (0.0146)
  MMP9 | -0.0017 (0.0100) | -0.0021 (0.0233)
  Total Protease | -22351.6 (102888.2) | -22540.9 (66146.2)

3. Secondary Outcome: Investigator's Global Assessment (IGA) Scores at Week 12
Description: Number of participants in each category of the Investigator's Global Assessment (IGA) scores at week 12. Investigator's Global Assessment evaluates papules and pustules of rosacea on a scale from 0 - 4 (0 = Clear, 1 = Near Clear, 2 = Mild, 3 = Moderate and 4 = Severe) with 0 being best and 4 being worst.
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Oracea® | Placebo
Number analyzed (Participants) | 84 | 86
participants
  Clear | 8 | 2
  Near Clear | 23 | 18
  Mild | 35 | 31
  Moderate | 12 | 20
  Severe | 6 | 15

4. Secondary Outcome: Change From Baseline in Clinician's Erythema Assessment (CEA) Scores
Description: Mean change in Clinician's Erythema Assessment (CEA) from baseline to week 12. Clinician's Erythema Assessment evaluates erythema on a scale from 0 - 4 (0 = None, 1 = Mild, 2 = Moderate, 3 = Significant and 4 = Severe) with 0 being best and 4 being worst.
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oracea® | Placebo
Number analyzed (Participants) | 84 | 86
units on a scale | -1.0 (2.9) | -0.8 (3.1)

ADVERSE EVENTS:
Arm/Group | Oracea® | Placebo
Serious Adverse Events (participants affected / at risk) | 2/84 | 0/86
Other Adverse Events (participants affected / at risk) | 8/84 | 6/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oracea® (N=84) | Placebo (N=86)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) — unlikely related to study drug
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oracea® (N=84) | Placebo (N=86)
nausea (Gastrointestinal disorders) | 3 (4) | 1 (2)
sinusitis (Infections and infestations) | 3 (3) | 2 (2)
upper respiratory infection (Infections and infestations) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days